CLINICAL TRIAL: NCT05478785
Title: A Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Efficacy of Cisplatin Micelle Injection (HA132) in Patients With Advanced Malignant Solid Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Efficacy of Cisplatin Micelle Injection (HA132) in Patients With Advanced Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HA132C-01
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Advanced Malignant Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cisplatin micelle injection (HA132) (Experimental): Dose-escalation: Five dose levels have been selected for evaluation in the Phase Ⅰ of the study. Dose escalation decisions will be determined based on toxicities observed during the first cycle.
  Dose-expansion: Patients will be administered HA132 at one or two dose levels (e.g. MTD and the dose below MTD).
  Cohort-expansion: Patients will be administered HA132 at one or two dose levels (e.g. MTD and the dose below MTD).
  Interventions: Drug: Cisplatin micelle injection (HA132)

INTERVENTIONS:
Drug: Cisplatin micelle injection (HA132) — HA132 will be administered intravenously (IV), once per 3 weeks.

SUMMARY:
This is a multicenter, open-label, dose-escalation, dose-expansion, and cohort-expansion Phase I/II clinical study to evaluate safety, tolerability, pharmacokinetics, antitumor efficacy and to determine the maximum tolerated dose (MTD) and recommended Phase 2 doses (RP2D) of cisplatin micelle injection in patients with advanced malignant solid tumors. This study is divided into two stages, the first stage (stage I) is the dose escalation and dose expansion study of cisplatin micelle injection, to determine the maximum tolerated dose (MTD), and to initially explore the recommended dose of phase II clinical practice (RP2D). The second stage (stage II) is the cisplatin micelle injection cohort expansion study to evaluate the efficacy and safety of cisplatin micelle injection (HA132) in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years (inclusive), no gender limitation;
2. Stage I: patients with advanced, recurrent or metastatic solid tumors confirmed by histology or cytology, and no standard treatment, or ineffective or intolerable to standard treatment, or those who are not eligible to receive standard treatment; Stage II: Pending;
3. Have at least one measurable lesion according to RECIST v1.1;
4. Eastern Cooperative Oncology Group (ECOG) physical performance status score of 0-1;
5. Life expectancy of at least 3 months;
6. Major organ function within 7 days prior to treatment, meeting the following criteria (have not received blood transfusion, EPO, G-CSF or other medical supportive treatment within 14 days before study drug administration):

   1. Blood routine:

      1. Neutrophil absolute value (ANC) ≥ 1.5 × 10^9/L;
      2. Platelet (PLT) ≥ 90× 10^9/L;
      3. Hemoglobin (HB) ≥ 90 g/L;
   2. Renal function:

      1. Creatinine (Cr) ≤ 1.5 × ULN;
      2. Creatinine clearance (CrcL) ≥ 60 mL/min (Using the Cockcroft-Gault formula);
   3. Liver function:

      1. Total bilirubin (TBIL) ≤ 1.5 × ULN;
      2. Aspartate amino transferase( AST) and Alanine amino transferase (ALT) 2.5 × ULN, or ≤ 5 × ULN in patients with hepatic metastasis or primary liver cancer;
      3. Alkaline phosphatase (ALP) ≤ 2.5 ×ULN, or ≤ 5 × ULN in patients with hepatic metastasis or primary liver cancer;
7. Women of childbearing age should agree that contraceptive measures (such as intrauterine device or condoms) must be used within study period and within 6 months after the end of the study; the serum or urine pregnancy tests is negative within 7days prior to the study for non-lactating patients; men should agree to use contraceptive measures during the study period and within 6 months after the end of the study period;
8. Patients must give informed consent to this study before the trial, and voluntarily sign the written informed consent.

Exclusion Criteria:

1. The patient has received chemotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy and other anti-tumor treatments or participated in other clinical trials within 4 weeks before the first use of the study drug, or within 5 half-lives of the treatment drug, whichever is longer;
2. The patient has received platinum-based therapy within 3 months prior to the study drug;
3. The patient has undergone major organ surgery (excluding needle biopsy) or suffered significant trauma within 4 weeks before the first use of the study drug;
4. The patient has received nephrotoxic or ototoxic drugs such as cephalosporin, aminoglycoside antibiotics, amphotericin B within 14 days before the first use of the study drug;
5. Those who are allergic to any excipients of the study drug or cisplatin and other platinum-based drug or have a history of severe allergies;
6. Any unresolved toxicities from prior anti-tumor therapy (including radiotherapy) greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1(except for alopecia or other adverse reactions judged no safety risk by the investigators);
7. Patients with clinical symptoms of central nervous system metastases or meningeal metastases, or there is other evidence that the patient's central nervous system metastases or meningeal metastases have not been controlled, and the investigators judge that they are not suitable for enrollment;
8. The patient has active infectious disease;
9. The patient has a history of autoimmune disease, immunodeficiency, including positive HIV test, or has other acquired, congenital immunodeficiency diseases, or a history of organ transplantation;
10. Active hepatitis B (hepatitis B virus titer > 1000 copies/mL or 200 IU/mL), prophylactic antiviral therapy other than interferon is allowed; hepatitis C virus infection;
11. Patients with a history of severe cardiovascular disease, or severe renal dysfunction, bone marrow insufficiency, chickenpox, herpes zoster, gout, hyperuricemia, or a history of other serious systemic diseases, as judged by the investigator who are not suitable to participate in clinical trials;
12. Known alcohol or drug dependence;
13. Patients with ototoxicity (except high-frequency elderly hearing loss) or other neurotoxicity ≥ grade 2 assessed by audiometer;
14. Patients with known visual impairment who are deemed unsuitable for participation in this study by the investigator;
15. Previous history of clear neurological or psychiatric disorders, including epilepsy or dementia;
16. Pregnant or breastfeeding females;
17. Patients with history of other malignancies within 3 years before the first use of the investigational drug, except for the following: cured basal cell or squamous cell skin cancer, superficial bladder cancer, prostate cancer in situ, cervical cancer in situ, breast cancer in situ, etc. locally curable cancer, or persistent disease-free survival within 3 years;
18. The investigator believes that the patients are not suitable to participate in this clinical study for other reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-limiting Toxicities (DLTs) in Stage I | Day 1 to 21 of Cycle 1 (each cycle of 21 days).
Incidence of adverse events in Stage I | From Baseline (Day 1) up to 28 days post last dose.
  Patients will be assessed for incidence and severity of adverse events(AEs) according to NCI-CTCAE criteria.
Maximum tolerated dose (MTD) in Stage I | Day 1 to 21 of Cycle 1 (each cycle of 21 days).
Recommended phase 2 dose (RP2D) in Stage I | Day 1 to 21 of Cycle 1 (each cycle of 21 days).
  The RP2D will be determined based on safety data including DLT, preliminary efficacy data,and PK data.
Objective Response Rate (ORR) in stage Ⅱ | Up to approximately 2 years.
  Proportion of patients whose best overall response is CR or PR in studies assessed according to RECIST v1.1.
Confirmed objective response rate (ORR) in stage Ⅱ | Up to approximately 2 years.
  During the study period, the best overall response is the proportion of patients with confirmed CR or PR (ie, CR+PR) as assessed by Response Evaluation Criteria in Solid Tumors.(RECIST v1.1).

SECONDARY OUTCOMES:
PK Indicator: Area under plasma concentration vs time curve(AUC)、Peak plasma concentration(Cmax)、Terminal Half Life（T1/2）. | Day 1 of Cycle 1 up to Day 1 of Last Cycle.
ORR in Stage I | Up to approximately 2 years.
Confirmed ORR in Stage I | Up to approximately 2 years.
Progression-free survival (PFS) | Up to approximately 2 years.
  Progression-free survival is defined as the time from the patient's first dose of study treatment (HA132) to the first date of either disease progression or death, whichever occurs first.
Disease control rate (DCR) | Up to approximately 2 years.
  Proportion of patients whose best overall response is CR, PR or SD in studies assessed according to RECIST v1.1.
Duration of response (DOR) | Up to approximately 2 years.
  The DOR for a responder is defined as the time from the patient's initial objective response to the first date of either disease progression or death, whichever occurs first.
Incidence of Adverse Events and Serious Adverse Events (SAEs) in stage Ⅱ | Up to approximately 2 years.
Estimated glomerular filtration rate (eGFR) and creatinine clearance | Up to approximately 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin Cancer Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No